CLINICAL TRIAL: NCT02525952
Title: A Randomized Controlled Trial to Compare the Outcomes Between Hepatectomy and Transarterial Chemoembolization for Patients With Multiple Hepatocellular Carcinomas Based on the NDR Scoring System
Brief Title: Treatment for Patients With Multiple Hepatocellular Carcinomas Based on the NDR Scoring System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHBHKY2015-01-012
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Carcinoma, Hepatocellular; Hepatectomy; Transarterial Chemoembolization; Scoring System
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Hepatectomy with NDR 0-2 (Experimental): Surgical removal of all lesions for patients with a NDR score 0-2 according to the NDR scoring system
  Interventions: Procedure: Hepatectomy
- TACE with NDR 0-2 (Active Comparator): Transarterial chemoembolization for patients with a NDR score 0-2 according to the NDR scoring system
  Interventions: Procedure: TACE
- Hepatectomy with NDR >2 (Experimental): Surgical removal of all lesions for patients with a NDR score more than 2 according to the NDR scoring system
  Interventions: Procedure: Hepatectomy
- TACE with NDR >2 (Active Comparator): Transarterial chemoembolization for patients with a NDR score more than 2 according to the NDR scoring system
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: Hepatectomy — Surgical removal of all lesions
  Arms: Hepatectomy with NDR 0-2; Hepatectomy with NDR >2
Procedure: TACE — Transarterial chemoembolization with lipiodol and pirarubicin
  Arms: TACE with NDR 0-2; TACE with NDR >2

SUMMARY:
The aim of this study is to establish a selection criteria of hepatectomy for patients with multiple hepatocellular carcinomas based on the NDR Scoring System

DETAILED DESCRIPTION:
Multiple hepatocellular carcinomas (HCCs) accounts for 60% to 70% of patients with hepatocellular carcinoma.However,the selection criteria of hepatectomy for patients with multiple HCCs remains controversial.Researches have suggested that part of the patients with multiple HCCs can also benefit from hepatectomy.But,expanding the selection criteria for hepatectomy will increase tumor recurrence rates and reduce the therapeutic effect, more stringent selection criteria will also make part of the patients who should take hepatectomy lose the operation chance. This is a difficult problem in the research of this field.The Barcelona Clinic Liver Cancer (BCLC) system recommends that stage A (number ≤ 3, largest diameter ≤ 3 cm) were suitable for liver resection.However, increasing reports on good outcome after hepatectomy for patients with multiple HCCs have been published.Studies on clonal origin suggest that hepatectomy is a better treatment for multiple HCCs from multicentric origin (MO) than that from intrahepatic metastasis (IM) and the 5-year overall survival rates is 24% to 58%.The investigators established a scoring system(NDR score; N, tumor number; D, total tumor diameter; R, ratio of largest/smallest diameter) based on preoperative data which can accurately predict postoperative long-term survival of patients with multiple HCCs.The formula is as follows: 1×N（N: >3=1; ≤3= 0）+ 2×D（D: >8cm = 1; ≤8cm= 0）+ 1×R（R: >6 = 1; ≤6= 0）.The investigators first propose a selection criteria of hepatectomy for patients with multiple HCCs based on this scoring system. Patients with a NDR score 0-2 are recommended for hepatectomy and can benefit from the surgery,and because of the unsatisfied outcome,patients with a NDR score more than 2 are not recommended for hepatectomy.The stringent selection criteria should be expanded so that more patients can benefit from hepatectomy,and the less stringent criteria should be limited to ensure curative effect.So,the investigators' NDR scoring system was more accurate in selecting patients with multiple HCCs for hepatectomy and this article was published on Ann Surg Oncol（2015，22:826）.In order to further confirm the rationality of this selection criteria,the investigators would like to propose a prospective randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years and <=70 years of age
2. Patients preoperatively diagnosed of hepatocellular carcinoma according to the criteria of American Association for the Study of Liver Diseases(AASLD).
3. Preoperative ECOG criteria score of 0-1
4. Child-Pugh class A liver function
5. Multiple hepatocellular carcinomas with tumor number <=5 and total tumor diameter <=15 cm

Exclusion Criteria:

1. Major portal/hepatic vein invasion
2. Extrahepatic metastasis
3. Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction,which may affect the treatment of liver cancer
4. Anticancer treatment before surgery
5. Lost to follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years

SECONDARY OUTCOMES:
Time to recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Feng, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China